CLINICAL TRIAL: NCT03020524
Title: A Pilot Study to Evaluate the Safety and Tolerability of Escalating Doses of Autologous CD4 T-Cells Modified With Lentiviral Vector Expressing an HR2, C34-peptide Conjugated to the CXCR4 N-terminus in HIV-infected Subjects
Brief Title: Autologous CD4 T-Cells in HIV (C34-CXCR4)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 826035
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

ARMS (3):
- Dose level 1: (Experimental): Autologous CD4 T-Cells0.8-1x10^9 transduced CD4+T-cells administered IV as a single dose
  Interventions: Biological: Autologous CD4 T-Cells
- Dose level 2 (Active Comparator): Autologous CD4 T-Cells 2.4-3x10^9 transduced CD4+ T-cells administered IV as a single dose
  Interventions: Biological: Autologous CD4 T-Cells
- Dose level 3 (Active Comparator): Autologous CD4 T-Cells 0.8-1x10^10 transduced CD4+ T-cells administered IV as a single dose
  Interventions: Biological: Autologous CD4 T-Cells

INTERVENTIONS:
Biological: Autologous CD4 T-Cells — all participants will receive a single infusion of C34-CXCR4-modified CD4+ T-cells at one of 3 dose levels. The first 3 subjects will receive dose level 1 of 0.8-1x109 transduced CD4+T-cells. Provided no dose limiting toxicity (DLT) is seen at the first dose level, the next 3 subjects will receive infusion at the 2nd dose level of 2.4-3x109 transduced CD4+ T-cells. If no DLT occurs at that dose, the final 3 subjects will receive the 3rd dose level of 0.8-1x1010 transduced CD4+ T-cells. In the event of a DLT (grade 3 or higher unexpected, related AE) recruitment will be paused pending DSMB decision

SUMMARY:
A single cohort, open-label pilot study of the safety and tolerability of a single infusion of autologous CD4+ T-cells genetically modified with an HR2, C34-peptide conjugated to the CXCR4 N-terminus using a lentiviral vector in HIV-infected subjects. This is a first in human study of C34-CXCR4 T cells

DETAILED DESCRIPTION:
There will be a single cohort in this study, which consists of subjects with well-controlled HIV replication on HAART. Within this cohort will be 3 escalating doses of T-cell infusions. A modified 3+3+3 dose-escalation design will be followed, in which the standard dose-escalation algorithm is stopped when a maximum of 9 evaluable subjects or a DLT stopping point has been reached, whichever comes first. At each dose level, three patients are treated. For dose levels 1 and 2, if 0/3 subjects have a dose limiting toxicity (DLT), then the dose is escalated. If 1/3 has a DLT (grade 3 or higher unexpected, related adverse event [AE]) at a dose level then 3 additional patients are treated at that dosage before escalating, and if <2/6 have DLT (i.e. no additional DLT is observed) then the dose is escalated to the next planned dose level and patients treated until a maximum of 9 evaluable subjects has been reached. The study will comprise of 5 steps:

Step 1, all participants will undergo leukapheresis to obtain CD4 positive T-cells that will be genetically modified. A second leukapheresis and a rectal biopsy will provide baseline specimens to evaluate the size of the HIV reservoir

Step 2, all participants will receive a single infusion of C34-CXCR4-modified CD4+ T-cells at one of 3 dose levels. The first 3 subjects will receive dose level 1 of 0.8-1x109 transduced CD4+T-cells. Provided no dose limiting toxicity (DLT) is seen at the first dose level, the next 3 subjects will receive infusion at the 2nd dose level of 2.4-3x109 transduced CD4+ T-cells. If no DLT occurs at that dose, the final 3 subjects will receive the 3rd dose level of 0.8-1x1010 transduced CD4+ T-cells. In the event of a DLT (grade 3 or higher unexpected, related AE) recruitment will be paused pending DSMB decision.

Step 3 all participants will participate in a 16-week analytical treatment interruption beginning 4 weeks after T-cell infusion.

At the end of step 3 all participants will undergo mini-leukapheresis and rectal biopsy

Step 4 all participants will be advised to resume antiretroviral therapy and will be followed until plasma HIV RNA falls below the limit of detection.

In Step 5 all participants will undergo leukapheresis and rectal biopsy at 52 weeks post infusion. At the completion of the study, participants will be asked to participate in a long-term follow-up study as required by regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to enrollment and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA VL.
* Ability and willingness of subject to provide informed consent.
* Men and women ages ≥18 years.
* Clinically stable on their first or second HAART regimen. Changes while the patient HIV viral load is undetectable does not count toward the number of ART regimens used, only changes made for virologic failure (for example an individual switching from an NNRTI-based regimen to an integrase inhibitor based regimen while the HIV viral load is undetectable will still be in their first regimen). Site investigator anticipates that a fully active alternative ART regimen could be constructed in the event of virologic failure on the current ART regimen.The current regimen should have no changes within 4 weeks of enrollment. Subjects must be willing to continue on current antiretroviral therapy for the duration of the study except for the duration of the 16 week analytical treatment interruption. (NOTE: changes to safely begin the treatment interruption are permitted).
* Screening HIV-1 RNA that is ≤50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 30 days prior to enrollment.
* HIV-1 RNA ≤50 copies/mL using a FDA-approved assay for at least 24 weeks prior to enrollment performed by any laboratory that has a CLIA certification or its equivalent.

  * NOTE: HIV-RNA must be measured at least once in the last 24 weeks and at least 3 days before the screening measure. Single determinations that are between >50 and <400 copies/mL (ie, blips) are allowed as long as the preceding and subsequent determinations are ≤50 copies/mL. The screening value may serve as the subsequent determination ≤50 copies/mL following a blip
  * NOTE: subjects who have participated in other trials using ATI's will be permitted since detectable virus during the interruption does not represent virologic failure. These subjects should have at least 24 weeks of VL <50 copies/mL.
* Screening CD4+ T-cell count ≥450 cells/ mm3 within 30 days of enrollment.
* Started ART with nadir CD4+ ≥200 cells/ mm3.
* The following laboratory values obtained within 30 days prior to enrollment meeting the following criteria:

  * Absolute neutrophil count (ANC) ≥1000 cells/mm3
  * Hemoglobin:≥10.0(males); ≥9.5 (females) g/dL
  * Platelet count: 100,000/mm3
  * Calculated creatinine clearance ≥50 mL/min estimated by the Cockcroft-Gault equation
  * Alanine aminotransferase (ALT) ≤ 2.0 x ULN
* Negative HBsAg within 6 months prior to enrollment.
* Negative HCV serology, or if positive, negative HCV RNA within 6 months prior to enrollment
* Adequate venous access and no other contraindications for leukapheresis.
* Have a Karnofsky Performance Score of 70 or higher.
* Have a recorded viral load set point prior to starting antiretroviral therapy

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection
* Current or prior AIDS diagnosis.
* History of cancer or malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin
* History or any features on physical examination indicative of active or unstable cardiac disease or hemodynamic instability.

  * NOTE: Subjects with a history of cardiac disease may participate with a physician's approval.
* History or any features on physical examination indicative of a bleeding diathesis
* Have been previously treated with any HIV experimental vaccine within 6 months prior to enrollment, or any previous gene therapy using an integrating vector.

  * NOTE: Subjects treated with placebo in an HIV vaccine study will not be excluded if documentation that they received placebo is provided.
* Use of chronic systemic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to enrollment.

  * NOTE: Recent or current use of inhaled steroids is not exclusionary. If subjects are prescribed a brief course of oral corticosteroids, the use should be limited to less than 7 days. Use of steroids before apheresis and immune assessment blood draws should be discouraged as it will affect white blood cell function.
* Breast-feeding, pregnant, or unwilling to use acceptable methods of birth control.
* Anticipated use of aspirin, dipyridamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2-week period prior to leukapheresis
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to enrollment
* Asymptomatic baseline serum chemistry elevations in LFTs, bilirubin, and serum creatinine due to HAART medication are not exclusionary, when in the opinion of the investigator, the abnormalities are not attributable to intrinsic hepatorenal disease. Such baseline elevations must be due to HAART.
* Receipt of vaccination within 30 days prior to enrollment.

  * NOTE: It is recommended that subjects enrolling into this study should have completed their routine vaccinations (hepatitis A, hepatitis B, pneumococcus, and tetanus diphtheria booster) at least 30 days prior to enrollment
* Have an allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennaylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Autologous CD4 T-Cells0.8-1x10^9 transduced CD4+T-cells administered IV as a single dose
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.9) | 40.7 (5.5) | 33.3 (10.2) | 37.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 1 | 2 | 1 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Treatment Related Adverse Events
Description: assessed by DAIDS AE grading table v2.0 November 2014
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 3 | 3
Participants | 2 | 1 | 2

2. Secondary Outcome: Compare the Percentage of Enriched Modified Cells C34-CXCR4 Modifiec T- Cells
Time Frame: 2 weeks post infusion, prior to ARV reinitiation, weeks 12, 16 and 20
Reporting Status: Not Posted

3. Secondary Outcome: Compare the Change Between CD4 Count
Time Frame: Baseline, week 2 post infusion, prior to ARV initiation, weeks 12, 16 20
Reporting Status: Not Posted

4. Secondary Outcome: Compare Viral Set Point Log 10 HIV RNA Level
Time Frame: week 2 post infusion, prior to ARV initiation, week 12, 16, 20
Reporting Status: Not Posted

5. Secondary Outcome: Evaluate Cell Mediated Response (Immunogenicity) Using Flow Cytometry
Time Frame: baseline through 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One year - Adverse events were collected from the time of informed consent to the completion of the scheduled study visits following the administration of study treatment.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3)
lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 1 | 2
rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 1
chills (General disorders) | 0 | 1 | 1
edema limbs (General disorders) | 1 | 0 | 0
fatigue (General disorders) | 2 | 2 | 0
pain (General disorders) | 0 | 1 | 0
vaccination site lymphadenopathy (General disorders) | 0 | 1 | 3
abscess (Infections and infestations) | 0 | 1 | 0
bronchial infection (Infections and infestations) | 0 | 1 | 0
gum infection (Infections and infestations) | 1 | 0 | 0
lymph gland infection (Infections and infestations) | 1 | 0 | 0
penile infection (Infections and infestations) | 1 | 1 | 0
pyuria (Infections and infestations) | 0 | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0
headache (Nervous system disorders) | 1 | 0 | 0
paresthesia (Nervous system disorders) | 0 | 0 | 1
strange smell sensation (Nervous system disorders) | 2 | 1 | 0
dysuria (Renal and urinary disorders) | 0 | 0 | 1
testicular mass (Reproductive system and breast disorders) | 0 | 1 | 0
vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
skin rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
tooth extraction (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03020524/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03020524/ICF_001.pdf